CLINICAL TRIAL: NCT03921346
Title: A Mobile Device App to Reduce Prehospital Medication Errors and Time to Drug Preparation and Delivery by EMS During Simulated Pediatric Cardiopulmonary Resuscitation: a Multicenter, Prospective, Randomized, Controlled Trial
Brief Title: Reducing Prehospital Medication Errors & Time to Drug Delivery by EMS During Simulated Pediatric CPR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pediatric Clinical Research Platform (Other)
Collaborators: University Hospital, Geneva (Other); University of Lausanne Hospitals (Other); Schutz & Rettung Sanitat (Other); Salva Servizio Ambulanza Locarnese e Valli (Other); Fribourg Emergency Medical Services, Fribourg, Switzerland (Other); Réseau Hospitalier Neuchâtelois (Other); Morges & Aubonne Emergency Medical Services (CSUMA), Morges and Aubonne, Switzerland (Other)
Responsible Party: Principal Investigator, Johan Siebert, MD, MD: Deputy Head, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SNSF_32003B_182374
Record Dates: First submitted 2019-04-12; First posted 2019-04-19 (Actual); Results first posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-06

CONDITIONS: Cardiopulmonary Arrest; Resuscitation; Pediatrics; Medication Errors; Emergency Medical Services
Keywords: Medication errors; Drugs; Pediatrics; Biomedical Technology; Mobile applications; Emergency Medical Services
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, randomized, controlled trial
Who Masked: Participant
Masking Description: Blinding to the direct IV drugs and doses intended for use will be maintained during recruitment to minimize preparation bias. Allocation concealment will be ensured with an allocation software and not released until the paramedics start the scenario. Study team members will be revealed to the participants just before the scenario starts. Paramedics will be unblinded when the simulated scenario starts. Although the intervention could not be masked, all investigators will remain unaware of the outcomes until all data will be unlocked for analysis at the end of the trial. All scenarios will be video-recorded for later analysis. Post-scenario video review will be done without blinding by two reviewers, but undertaken independently and blinded to each other's reviews. In case of disagreement, a third independent evaluator will help reach a consensus. The data analyst will be blinded to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (mobile device app) (Experimental): Paramedics preparing drugs with the help of the mobile device app PedAMINES™.
  Each paramedic will have to prepare sequentially 4 direct IV emergency drugs with the help of the mobile device app PedAMINES™.
  Interventions: Device: Mobile device app (PedAMINES™) 1st drug; Device: Mobile device app (PedAMINES™) 2nd drug; Device: Mobile device app (PedAMINES™) 3rd drug; Device: Mobile device app (PedAMINES™) 4th drug
- Arm B (conventional preparation method) (Active Comparator): Paramedics preparing drugs with the help of conventional method.
  Each paramedic will have to prepare sequentially 4 direct IV emergency drugs with the help of conventional method
  Interventions: Device: Conventional method 1st drug; Device: Conventional method 2nd drug; Device: Conventional method 3rd drug; Device: Conventional method 4th drug

INTERVENTIONS:
Device: Mobile device app (PedAMINES™) 1st drug — To prepare 0.01 mg/kg epinephrine (0.1 mL/kg of 0.1 mg/mL concentration)
  Arms: Arm A (mobile device app)
Device: Mobile device app (PedAMINES™) 2nd drug — To prepare 0.1 mg/kg midazolam (of 5 mg/mL concentration ad 10 mL sodium chloride 0.9%)
  Arms: Arm A (mobile device app)
Device: Mobile device app (PedAMINES™) 3rd drug — To prepare 4 mL/kg dextrose 10%
  Arms: Arm A (mobile device app)
Device: Mobile device app (PedAMINES™) 4th drug — To prepare 1 mmol/kg sodium bicarbonate (of 4.2% = 0.5 mmol/L concentration)
  Arms: Arm A (mobile device app)
Device: Conventional method 1st drug — To prepare 0.01 mg/kg epinephrine (0.1 mL/kg of 0.1 mg/mL concentration)
  Arms: Arm B (conventional preparation method)
Device: Conventional method 2nd drug — To prepare 0.1 mg/kg midazolam (of 5 mg/mL concentration ad 10 mL sodium chloride 0.9%)
  Arms: Arm B (conventional preparation method)
Device: Conventional method 3rd drug — To prepare 4 mL/kg dextrose 10%
  Arms: Arm B (conventional preparation method)
Device: Conventional method 4th drug — To prepare 1 mmol/kg sodium bicarbonate (of 4.2% = 0.5 mmol/L concentration)
  Arms: Arm B (conventional preparation method)

SUMMARY:
The study investigators will recruit paramedics in many Emergency Medical Services (EMS) in Switzerland to prepare direct intravenous (IV) emergency drugs during a standardized simulation-based pediatric out-of-hospital cardiac arrest scenario. According to randomization, each paramedic will be asked to prepare sequentially 4 IV emergency drugs (epinephrine, midazolam, dextrose 10%, sodium bicarbonate 4.2%) following either their current conventional methods or by the aim of a mobile device app. This app is designed to support drug preparation at pediatric dosages. In a previous multicenter randomized trial with nurses, the investigators reported the ability of this app to significantly reduce in-hospital continuous infusion medication error rates and drug preparation time compared to conventional preparation methods during simulation-based resuscitations. In this trial, the aim was to assess this app during pediatric out-of-hospital cardiopulmonary resuscitation with paramedics.

DETAILED DESCRIPTION:
Children represent a vulnerable population with specific medical needs compared to adults. Fast, accurate, and safe preparation and administration of IV drugs is both complex and time consuming in pediatric critical situations, such as cardiopulmonary resuscitation (CPR). Most drugs given IV to children are provided in vials originally prepared for the adult population, which leads to the need for a specific individual, weight-based drug dose calculation and preparation for each child that varies widely across age groups. This error-prone process and the lower dosing error tolerance of children place them at a high risk for life-threatening medication errors. Despite well equipped and staffed environments with numerous available safeguards, direct IV medication errors have been reported in up to 41% of cases during simulated in-hospital pediatric resuscitations, 65% of which were incorrect medication dosage, making it the most common error. The rate of errors is also important in the prehospital setting, occurring in more than 30% of all pediatric drugs administered. As paramedics have little exposure to critically ill children, they have limited opportunities to administer resuscitation drugs at pediatric doses and to train this skill.

Moreover, in resuscitation, time is inversely correlated to survival. During the first 15 min of in-hospital pediatric CPR, survival and favorable neurological outcome decrease linearly by 2,1% and 1,2% per min, respectively, and rely in part on drug preparation time either in- or out-of-hospital. Among non-shockable pediatric out-of-hospital cardiac arrests, each minute delay to epinephrine delivery is associated with 9% decrease in the odds of survival. Regrettably, in the prehospital setting, the majority of patients receive epinephrine more than 10 minutes after EMS arrival. The chain of survival therefore critically relies on early out-of-hospital CPR by EMS, and onsite administration of IV emergency drugs without delay before a rapid transfer to pediatric emergency departments and advanced care.

In a previous multicenter, randomized crossover trial, medication errors, time to drug preparation, and time to drug delivery for continuous infusions during simulation-based pediatric in-hospital postcardiac arrest scenarios were significantly reduced by using a mobile device app - the pediatric accurate medication in emergency situations (PedAMINES™) app - designed to help pediatric drug preparation.

The present multicenter trial aims to compare the impact of this app with conventional calculation methods for the preparation of direct IV drugs during standardized, simulation-based, pediatric out-of-hospital cardiac arrest scenarios. The investigators hypothesized that use of the app might extend and scale up the previous multicenter in-hospital observations by similarly reducing occurrence of medication errors and time to drug preparation and delivery when used by paramedics in out-of-hospital settings.

In this trial, the investigators will recruit paramedics in many EMS in Switzerland to prepare direct IV emergency drugs during a standardized simulation-based pediatric out-of-hospital cardiac arrest scenario with a high-fidelity WiFi manikin (Laerdal SimBaby). The scenario will take place out-of-hospital in a simulated children's room to increase realism.

On the day of participation after random allocation (1:1 allocation ratio), each participating paramedic will (1) complete a survey collecting data regarding their demographics, care training, and simulation and computer experience, (2) receive a standardized 5-min training session on how to use the app, and (3) be presented the simulation manikin characteristics. The paramedics will then be asked to perform a 20-min highly realistic pediatric CPR scenario on the high-fidelity manikin. Each paramedic will be asked to prepare sequentially 4 intravenous emergency drugs (epinephrine, midazolam, dextrose 10%, sodium bicarbonate 4.2%) following either their current conventional methods or by the aim of the mobile app. The procedure is standardized across all sites to follow the same chronological progression and range of difficulty to ensure each participant is exposed to exactly the same case, with similar challenges in decision making and treatment preparation provided on the same manikin.

All the actions (i.e. primary and secondary outcomes) performed by the paramedics during the scenario will be automatically recorded and stored by the responsive simulator detectors, the app, and by several GoPro Hero 5 Black edition action video cameras worn by the paramedics and placed within the room.

The study will be carried out in accordance with the Consolidated Standards of Reporting Trials of Electronic and Mobile Health Applications and Online TeleHealth (CONSORT-EHEALTH) guidelines and the Reporting Guidelines for Health Care Simulation Research.

This study aims to compare the impact of this app with conventional calculation methods for the preparation of direct IV drugs during standardized, simulation-based, pediatric out-of-hospital cardiac arrest scenarios, were paramedics are little exposed to pediatric CPRs. The investigators hypothesize that use of the app might extend and scale up their previous multicenter in-hospital observations by similarly reducing occurrence of medication errors and time to drug preparation and delivery when used by paramedics in out-of-hospital settings.

ELIGIBILITY:
Inclusion Criteria:

* To be paramedic certified
* To know how to prepare direct IV drugs
* To have previously completed the 5-minute introductory course to the use of the app PedAMINES™ dispensed by the study investigators
* Participation agreement

Exclusion Criteria:

* To have at any time previously used the app PedAMINES™
* To have not undergone the 5-minute introductory course to the use of the app PedAMINES™

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johan N Siebert, MD, Principal Investigator — Geneva Children's Hospital, Geneva University Hospitals, Geneva, Switzerland
Locations (1):
- Geneva Emergency Medical Services (ACE Ambulances), Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
IPD will be deidentified and the study investigators will house the data locally on secure hard disk drives at the Geneva Children's Hospital. The datasets used or analyzed during the current trial will be available from the corresponding author upon reasonable request. Only deidentified/anonymized data will be shared.
Supporting Information: Study Protocol
Time Frame: Available from 1 month to 10 years after trial publication.
Access Criteria: From the corresponding author upon reasonable request.

REFERENCES:
- [Background] Siebert JN, Ehrler F, Combescure C, Lovis C, Haddad K, Hugon F, Luterbacher F, Lacroix L, Gervaix A, Manzano S; PedAMINES Trial Group. A mobile device application to reduce medication errors and time to drug delivery during simulated paediatric cardiopulmonary resuscitation: a multicentre, randomised, controlled, crossover trial. Lancet Child Adolesc Health. 2019 May;3(5):303-311. doi: 10.1016/S2352-4642(19)30003-3. Epub 2019 Feb 21. PMID 30797722
- [Background] Kaufmann J, Laschat M, Wappler F. Medication errors in pediatric emergencies: a systematic analysis. Dtsch Arztebl Int. 2012 Sep;109(38):609-16. doi: 10.3238/arztebl.2012.0609. Epub 2012 Sep 21. PMID 23093991
- [Background] Moreira ME, Hernandez C, Stevens AD, Jones S, Sande M, Blumen JR, Hopkins E, Bakes K, Haukoos JS. Color-Coded Prefilled Medication Syringes Decrease Time to Delivery and Dosing Error in Simulated Emergency Department Pediatric Resuscitations. Ann Emerg Med. 2015 Aug;66(2):97-106.e3. doi: 10.1016/j.annemergmed.2014.12.035. Epub 2015 Feb 18. PMID 25701295
- [Background] Kaushal R, Bates DW, Landrigan C, McKenna KJ, Clapp MD, Federico F, Goldmann DA. Medication errors and adverse drug events in pediatric inpatients. JAMA. 2001 Apr 25;285(16):2114-20. doi: 10.1001/jama.285.16.2114. PMID 11311101
- [Background] Hoyle JD, Davis AT, Putman KK, Trytko JA, Fales WD. Medication dosing errors in pediatric patients treated by emergency medical services. Prehosp Emerg Care. 2012 Jan-Mar;16(1):59-66. doi: 10.3109/10903127.2011.614043. Epub 2011 Oct 14. PMID 21999707
- [Background] Hoyle JD Jr, Crowe RP, Bentley MA, Beltran G, Fales W. Pediatric Prehospital Medication Dosing Errors: A National Survey of Paramedics. Prehosp Emerg Care. 2017 Mar-Apr;21(2):185-191. doi: 10.1080/10903127.2016.1227001. Epub 2017 Feb 8. PMID 28257249
- [Background] Porter E, Barcega B, Kim TY. Analysis of medication errors in simulated pediatric resuscitation by residents. West J Emerg Med. 2014 Jul;15(4):486-90. doi: 10.5811/westjem.2014.2.17922. PMID 25035756
- [Background] Shah MN, Cushman JT, Davis CO, Bazarian JJ, Auinger P, Friedman B. The epidemiology of emergency medical services use by children: an analysis of the National Hospital Ambulatory Medical Care Survey. Prehosp Emerg Care. 2008 Jul-Sep;12(3):269-76. doi: 10.1080/10903120802100167. PMID 18584491
- [Background] Su E, Schmidt TA, Mann NC, Zechnich AD. A randomized controlled trial to assess decay in acquired knowledge among paramedics completing a pediatric resuscitation course. Acad Emerg Med. 2000 Jul;7(7):779-86. doi: 10.1111/j.1553-2712.2000.tb02270.x. PMID 10917328
- [Background] Matos RI, Watson RS, Nadkarni VM, Huang HH, Berg RA, Meaney PA, Carroll CL, Berens RJ, Praestgaard A, Weissfeld L, Spinella PC; American Heart Association's Get With The Guidelines-Resuscitation (Formerly the National Registry of Cardiopulmonary Resuscitation) Investigators. Duration of cardiopulmonary resuscitation and illness category impact survival and neurologic outcomes for in-hospital pediatric cardiac arrests. Circulation. 2013 Jan 29;127(4):442-51. doi: 10.1161/CIRCULATIONAHA.112.125625. Epub 2013 Jan 22. PMID 23339874
- [Background] Andersen LW, Berg KM, Saindon BZ, Massaro JM, Raymond TT, Berg RA, Nadkarni VM, Donnino MW; American Heart Association Get With the Guidelines-Resuscitation Investigators. Time to Epinephrine and Survival After Pediatric In-Hospital Cardiac Arrest. JAMA. 2015 Aug 25;314(8):802-10. doi: 10.1001/jama.2015.9678. PMID 26305650
- [Background] Hansen M, Schmicker RH, Newgard CD, Grunau B, Scheuermeyer F, Cheskes S, Vithalani V, Alnaji F, Rea T, Idris AH, Herren H, Hutchison J, Austin M, Egan D, Daya M; Resuscitation Outcomes Consortium Investigators. Time to Epinephrine Administration and Survival From Nonshockable Out-of-Hospital Cardiac Arrest Among Children and Adults. Circulation. 2018 May 8;137(19):2032-2040. doi: 10.1161/CIRCULATIONAHA.117.033067. Epub 2018 Mar 6. PMID 29511001
- [Background] Fukuda T, Kondo Y, Hayashida K, Sekiguchi H, Kukita I. Time to epinephrine and survival after paediatric out-of-hospital cardiac arrest. Eur Heart J Cardiovasc Pharmacother. 2018 Jul 1;4(3):144-151. doi: 10.1093/ehjcvp/pvx023. PMID 29036580
- [Background] Foltin GL, Richmond N, Treiber M, Skomorowsky A, Galea S, Vlahov D, Blaney S, Kusick M, Silverman R, Tunik MG. Pediatric prehospital evaluation of NYC cardiac arrest survival (PHENYCS). Pediatr Emerg Care. 2012 Sep;28(9):864-8. doi: 10.1097/PEC.0b013e3182675e70. PMID 22929131
- [Background] Rittenberger JC, Bost JE, Menegazzi JJ. Time to give the first medication during resuscitation in out-of-hospital cardiac arrest. Resuscitation. 2006 Aug;70(2):201-6. doi: 10.1016/j.resuscitation.2005.12.006. Epub 2006 Jun 27. PMID 16806636
- [Background] Eysenbach G; CONSORT-EHEALTH Group. CONSORT-EHEALTH: improving and standardizing evaluation reports of Web-based and mobile health interventions. J Med Internet Res. 2011 Dec 31;13(4):e126. doi: 10.2196/jmir.1923. PMID 22209829
- [Background] Cheng A, Kessler D, Mackinnon R, Chang TP, Nadkarni VM, Hunt EA, Duval-Arnould J, Lin Y, Cook DA, Pusic M, Hui J, Moher D, Egger M, Auerbach M; International Network for Simulation-based Pediatric Innovation, Research, and Education (INSPIRE) Reporting Guidelines Investigators. Reporting Guidelines for Health Care Simulation Research: Extensions to the CONSORT and STROBE Statements. Simul Healthc. 2016 Aug;11(4):238-48. doi: 10.1097/SIH.0000000000000150. PMID 27465839
- [Background] Venkatesh, V., Morris, M. G., Davis, G. B., & Davis, F. D. (2003). User acceptance of information technology: Toward a unified view. MIS quarterly, 425-478.
- [Derived] Siebert JN, Gosetto L, Sauvage M, Bloudeau L, Suppan L, Rodieux F, Haddad K, Hugon F, Gervaix A, Lovis C, Combescure C, Manzano S, Ehrler F; PedAMINES Trial Group; PedAMINES Prehospital Group. Usability Testing and Technology Acceptance of an mHealth App at the Point of Care During Simulated Pediatric In- and Out-of-Hospital Cardiopulmonary Resuscitations: Study Nested Within 2 Multicenter Randomized Controlled Trials. JMIR Hum Factors. 2022 Mar 1;9(1):e35399. doi: 10.2196/35399. PMID 35230243
- [Derived] Lacour M, Bloudeau L, Combescure C, Haddad K, Hugon F, Suppan L, Rodieux F, Lovis C, Gervaix A, Ehrler F, Manzano S, Siebert JN; PedAMINES Prehospital Group. Impact of a Mobile App on Paramedics' Perceived and Physiologic Stress Response During Simulated Prehospital Pediatric Cardiopulmonary Resuscitation: Study Nested Within a Multicenter Randomized Controlled Trial. JMIR Mhealth Uhealth. 2021 Oct 7;9(10):e31748. doi: 10.2196/31748. PMID 34617916
- [Derived] Siebert JN, Bloudeau L, Combescure C, Haddad K, Hugon F, Suppan L, Rodieux F, Lovis C, Gervaix A, Ehrler F, Manzano S; Pediatric Accurate Medication in Emergency Situations (PedAMINES) Prehospital Group. Effect of a Mobile App on Prehospital Medication Errors During Simulated Pediatric Resuscitation: A Randomized Clinical Trial. JAMA Netw Open. 2021 Aug 2;4(8):e2123007. doi: 10.1001/jamanetworkopen.2021.23007. PMID 34459905
- [Derived] Siebert JN, Bloudeau L, Ehrler F, Combescure C, Haddad K, Hugon F, Suppan L, Rodieux F, Lovis C, Gervaix A, Manzano S. A mobile device app to reduce prehospital medication errors and time to drug preparation and delivery by emergency medical services during simulated pediatric cardiopulmonary resuscitation: study protocol of a multicenter, prospective, randomized controlled trial. Trials. 2019 Nov 20;20(1):634. doi: 10.1186/s13063-019-3726-4. PMID 31747951

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A (Mobile Device App): Paramedics preparing drugs with the help of the mobile device app PedAMINES™.
  Each paramedic will have to prepare sequentially 4 direct IV emergency drugs with the help of the mobile device app PedAMINES™.
  Mobile device app (PedAMINES™) 1st drug: To prepare 0.01 mg/kg epinephrine (0.1 mL/kg of 0.1 mg/mL concentration)
  Mobile device app (PedAMINES™) 2nd drug: To prepare 0.1 mg/kg midazolam (of 5 mg/mL concentration ad 10 mL sodium chloride 0.9%)
  Mobile device app (PedAMINES™) 3rd drug: To prepare 4 mL/kg dextrose 10%
  Mobile device app (PedAMINES™) 4th drug: To prepare 1 mmol/kg sodium bicarbonate (of 4.2% = 0.5 mmol/L concentration)
- Arm B (Conventional Preparation Method): Paramedics preparing drugs with the help of conventional method.
  Each paramedic will have to prepare sequentially 4 direct IV emergency drugs with the help of conventional method
  Conventional method 1st drug: To prepare 0.01 mg/kg epinephrine (0.1 mL/kg of 0.1 mg/mL concentration)
  Conventional method 2nd drug: To prepare 0.1 mg/kg midazolam (of 5 mg/mL concentration ad 10 mL sodium chloride 0.9%)
  Conventional method 3rd drug: To prepare 4 mL/kg dextrose 10%
  Conventional method 4th drug: To prepare 1 mmol/kg sodium bicarbonate (of 4.2% = 0.5 mmol/L concentration)
Period: Overall Study
Arm/Group | Arm A (Mobile Device App) | Arm B (Conventional Preparation Method)
Started | 74 | 76
Completed | 74 | 76
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Mobile Device App) | Arm B (Conventional Preparation Method) | Total
Number analyzed (Participants) | 74 | 76 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.7 (7.3) | 35.5 (7.1) | 35.6 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 23 | 49
  Male | 48 | 53 | 101
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Switzerland | 74 | 76 | 150
Proficiency in the use of smartphones or tablets (5-point Likert scale) [Count of Participants; unit: Participants]
  Strongly disagree | 1 | 0 | 1
  Disagree | 3 | 3 | 6
  Neutral | 12 | 13 | 25
  Agree | 38 | 48 | 86
  Strongly agree | 20 | 12 | 32
Time since paramedic certification (years, categorical) [Count of Participants; unit: Participants]
  <5 years | 26 | 27 | 53
  5 to10 years | 29 | 26 | 55
  >10 years | 19 | 23 | 42
Specific pediatric training (categorical) [Count of Participants; unit: Participants]
  Yes | 37 | 35 | 72
  No | 37 | 41 | 78
Time since last pediatric cardiopulmonary resuscitation (months, categorical) [Count of Participants; unit: Participants]
  Never | 32 | 30 | 62
  ≥24 | 26 | 28 | 54
  12 to <24 | 11 | 11 | 22
  6 to <12 | 4 | 5 | 9
  <6 | 1 | 2 | 3
Time since last preparation of emergency drugs (months, categorical) [Count of Participants; unit: Participants]
  Never | 9 | 12 | 21
  ≥24 | 18 | 18 | 36
  12 to <24 | 15 | 17 | 32
  6 to <12 | 17 | 7 | 24
  <6 | 15 | 22 | 37
Satisfaction with current drug preparation methods (5-point Likert scale) [Count of Participants; unit: Participants]
  Very unsatisfied | 9 | 8 | 17
  Unsatisfied | 18 | 19 | 37
  Neutral | 25 | 22 | 47
  Satisfied | 21 | 24 | 45
  Very satisfied | 1 | 3 | 4
Proficient with intravenous drug preparation (5-point Likert scale) [Count of Participants; unit: Participants]
  Strongly disagree | 9 | 7 | 16
  Disagree | 15 | 30 | 45
  Neutral | 30 | 14 | 44
  Agree | 19 | 22 | 41
  Strongly agree | 1 | 3 | 4
Attitude toward new technology (5-point Likert scale) [Count of Participants; unit: Participants]
  Strongly unfavorable | 0 | 0 | 0
  Unfavorable | 0 | 1 | 1
  Neutral | 6 | 1 | 7
  Favorable | 24 | 17 | 41
  Strongly favorable | 44 | 57 | 101

OUTCOME MEASURES:

1. Primary Outcome: Medication Dosage Errors
Description: To measure in each allocation group the number and percentage of medication dosage containing errors that occur during the sequence from drug preparation to drug injection. We define an emergency medication dose administration error as a failure in drug preparation if at least one of the following errors is committed: a deviation in drug dose of more than 10% from the correct weight dose; inability to calculate drug dosage without guidance help from the paramedic investigator (LB) leading the resuscitation in the room; and/or (because of its clinical relevance) a deviation of more than 10% of the final administered concentration of sodium bicarbonate from the prescribed 4.2% concentration. These errors will be measured both as the percentage deviation from the amount of delivered drug compared with the correct weight dose as prescribed by the physician and the absolute deviations from that dose.
Time Frame: 20 minutes
Measure: Mean (95% Confidence Interval); unit: percentage of medication errors
Arm/Group | Arm A (Mobile Device App) | Arm B (Conventional Preparation Method)
Number analyzed (Participants) | 74 | 76
percentage of medication errors | 5.7 [3.4 to 9.0] | 62.8 [57.1 to 68.3]

2. Secondary Outcome: Time to Drug Preparation and Time to Drug Delivery
Description: Secondary outcome will be the elapsed time in seconds between the oral prescription by the physician and a) time to drug preparation completion and b) time to drug delivery by the participant.
Time Frame: 20 minutes
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Arm A (Mobile Device App) | Arm B (Conventional Preparation Method)
Number analyzed (Participants) | 74 | 76
seconds
  Time to drug preparation | 146.6 [95.3 to 198.0] | 186.1 [134.8 to 237.4]
  Time to drug delivery | 186.8 [142.1 to 231.4] | 233.3 [188.7 to 277.9]

3. Secondary Outcome: Type of Medication Errors
Description: Incorrect preparations: a) drug dose deviation >10% from the correct dose prescribed by the physician, b) drug preparation necessitating assistance (i.e., inability for the nurse to prepare the prescribed drug without the help of a third party), and c) >10% deviation from the prescribed drug dose in the 4th drug concentration will be reported.
Time Frame: During each of the 4 drug preparations, an average of 20 minutes per drug preparation.
Population: Categories are not mutually exclusive. Various errors can occur during each drug preparation and therefore can be counted more than once
Measure: Count of Units; unit: Drug preparations
Units Other Than Participants: Drug preparations
Arm/Group | Arm A (Mobile Device App) | Arm B (Conventional Preparation Method)
Number analyzed (Participants) | 74 | 76
Number analyzed (Drug preparations) | 296 | 304
Drug preparations
  Incorrect preparations | 17 | 191
  Dose deviation >10% | 16 | 172
  Help required | 0 | 55
  4th drug concentration deviation >10% | 5 | 46

4. Secondary Outcome: Perceived Stress
Description: Participants' self-assessed psychological stress will be measured before and after the intervention (ie. drug preparation) using the Gauthier and Bouchard's French-Canadian adaptation of Spielberger's psychometric State-Trait Anxiety Inventory (STAI) Form Y-1 questionnaire. STAI ranges from 20 to 80, with higher scores being positively correlated with greater stress.
  Perceived stress will also be assessed by self-assessment using a numerical 10-point Likert visual analogue scale (VAS). Values range from 1 (totally unstressed) to 10 (totally stressed) to avoid neutral answers.
  The perceived stress before the preparation of the 4 drugs and after the preparation of the 4 drugs will be indicated for each study arm. In other words, the perceived stress will not be given for each of the 4 drugs individually, but as a single value before and a single value after the drug preparation, for both the STAI and the VAS.
Time Frame: At preintervention and postintervention, a total of 20 minutes will be used to complete the STAI questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Mobile App: Participants preparing the emergency drugs using the mobile app PedAMINES
- Conventional Method: Participants preparing the emergency drugs using conventional preparation methods
Arm/Group | Mobile App | Conventional Method
Number analyzed (Participants) | 73 | 76
score on a scale
  STAI preintervention | 36.1 (8.1) | 35.4 (8.2)
  STAI postintervention | 39.0 (8.4) | 49.8 (13.2)
  VAS preintervention | 4.2 (2.5) | 3.9 (2.2)
  VAS postintervention | 6.4 (1.9) | 7.1 (1.8)

5. Secondary Outcome: Stress Level Measured by Heart Rate Monitoring (Smartwatch).
Description: The participants' stress level will be assessed by measuring continuously their heart rate using a Polar A360 smartwatch on their wrist during the resuscitation scenario. Mean delta HR values (difference between HR peak values and baseline HR) will be obtained during some small segments of scenario and correlated to the scenario phases and the preparation methods used.
Time Frame: Baseline, recovery, and during each of the 4 drug preparations, a total of 20 minutes per participant will be used to continuously record heart rates on the smartwatch. Maximal HRpeak is the maximum HR across all preparations
Population: Outcome measures are expressed as mean [SD] beats per minute per study group (with no minimum nor maximum values as heart rates can vary greatly between individuals)
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Mobile App | Conventional Method
Number analyzed (Participants) | 73 | 76
Beats per minute
  Baseline heart rate (HR) | 79.3 (14.4) | 78.5 (12.7)
  First drug, HRpeak | 123.1 (9.2) | 124.1 (12.2)
  Second drug, HRpeak | 121.1 (10.9) | 119.9 (13.3)
  Third drug, HRpeak | 120.4 (11.4) | 117.9 (13.3)
  Fourth drug, HRpeak | 114.1 (13.5) | 110.5 (13.7)
  Recovery (directly after the intervention, at rest in the absence of drug preparation) | 79.3 (15.0) | 76.8 (13.7)
  Maximal HRpeak | 126.1 (10.3) | 126.0 (12.1)

6. Secondary Outcome: Unified Theory of Acceptance and Use of Technology (UTAUT) Questionnaire and System Usability Score (SUS)
Description: Unified Theory of Acceptance and Use of Technology (UTAUT): a 52-item questionnaire distributed in 8 core constructs: 1) perceived usefulness (4 items), 2) perceived ease of use (4 items), 3) task-technology fit (4 items), 4) performance expectancy (3 items), 5) impact on image (2 items), 6) personal innovativeness (3 items), 7) acceptance (3 items), and 8) behavioral intention to use the technology (3 items). Each construct are based on a Likert-type 5-point scale ranging from 1 (strongly disagree) to 5 (strongly agree). Increments are integers between 1 to 5. Min score per construct = 1, max score per construct = 5. The higher the score, the better the acceptance.
  System Usability Score (SUS): Comprises a 10-item questionnaire with 5 response options for each item, ranging from 1 (strongly disagree) to 5 (strongly agree). The higher the score, the better the usability (ie, 0=very poor perceived usability and 100=excellent perceived usability)
Time Frame: 60 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A (Mobile Device App)
Number analyzed (Participants) | 74
score on a scale
  Perceived usefulness - UTAUT | 4.69 (0.44)
  Perceived ease of use - UTAUT | 4.61 (0.35)
  Task-technology fit - UTAUT | 4.49 (0.54)
  Performance expectancy - UTAUT | 4.55 (0.59)
  Impact on image - UTAUT | 4.74 (0.57)
  Personal innovativeness - UTAUT | 4.14 (0.58)
  Acceptance - UTAUT | 4.32 (0.61)
  Behavioral intention to use the technology - UTAUT | 4.81 (0.34)
  SUS | 89.7 (8.7)

ADVERSE EVENTS:
Time Frame: 0
Description: As this simulation-based study will not involve patient enrollment and will not expose participants (i.e., paramedics) to risks beyond their routine clinical practice, no adverse events will be recorded nor monitored. A manikin will be used to run the CRP scenarios and not a real patient.
Arm/Group | Arm A (Mobile Device App) | Arm B (Conventional Preparation Method)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-29): https://cdn.clinicaltrials.gov/large-docs/46/NCT03921346/Prot_SAP_000.pdf